CLINICAL TRIAL: NCT00549432
Title: Clinical Study of Abdominal Aortic Aneurysm Exclusion Using the TALENT Enhanced LPS Endoluminal Stent-Graft System
Brief Title: Clinical Study of Abdominal Aortic Aneurysm Exclusion (TALENT Abdominal)
Acronym: l
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Edward B. Diethrich, MD, Arizona Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G020149
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: TALENT Enhanced LPS Endoluminal Stent-Graft System

INTERVENTIONS:
Device: TALENT Enhanced LPS Endoluminal Stent-Graft System — roadmapping, and angiography for proper implant positioning. The TALENT endoluminal stent-graft endoprosthesis is inserted by delivery catheter and introducer sheath via a surgical cutdown (e.g., external iliac artery, femoral artery) approach. The insertion method depends on each patient's anatomy and is determined by the Clinical Investigator.

SUMMARY:
The purpose of the study is to evaluate the TALENT endoluminal stent-graft system in patients with abdominal aortic aneurysms. The TALENT endoluminal stent-graft system is a flexible, implantable endoluminal vascular device preloaded in a placement system that is used to exclude abdominal aortic aneurysms.

DETAILED DESCRIPTION:
An aneurysm is a localized dilatation of a blood vessel at least 1 1/2 to 2 times the normal vessel diameter. Abdominal aortic aneurysms are relatively common, and have been detected in 1.3% to 2.7% of patients 65 to 80 years of age (Blum, et al, 1996; Collins, Araujo, and Lindsell, 1988; Scott, Ashton, and Kay, 1991). A large proportion (up to 50%) of patients with untreated AAAs experience rupture and exsanguination (Johansen, 1995). Ruptured AAAs are the 13th leading cause of death in the US, accounting for more than 15,000 deaths per year (Cronenwett and Sampson, 1995).

Conventional treatment of abdominal aortic aneurysms is by a surgical procedure involving midline laparotomy, aortic clamping, aortic bypass, and blood loss with associated transfusion. Improvements in surgical techniques and patient care have allowed the mortality rate associated with this procedure to be reduced to approximately 5%, when elective repair is done prior to rupture of the aneurysm. Risks of surgery increase when the patient is considered to be a poor candidate for surgery.

Due to progress made in interventional radiology and endovascular surgery, it is now possible to treat aneurysms without an abdominal surgical procedure, thus potentially further reducing the risks associated with elective repair. This new therapeutic approach consists of transfemoral introduction of a metallic stent coupled with a vascular graft. When the stent device is deployed and expanded within the aneurysmal blood vessel, it creates a new aortic lumen for blood flow, effectively excluding the aneurysm sac from the flow while maintaining perfusion to the lower limbs. This less invasive technique is designed to prevent the need for laparotomy, to reduce the need for blood transfusions, to decrease the use of anesthetics and other drugs, and to speed recovery time.

The objective of this study is to evaluate the safety and effectiveness of the TALENT endoluminal stent-graft system in patients who may be categorized as standard risk, high risk or other indications. Standard risk patients are patients with indications for treatment that are consistent with those for a manufacturer IDE, when there is no active enrollment in the IDE. High risk patients are patients who do not meet the entrance criteria for the manufacturer sponsored IDE as they are at high risk of morbidity and mortality with standard surgical repair. Other indications would be considered patients with indications for treatment outside of those or the manufacturer sponsored IDE.

This study will be performed in both high risk and low risk patients who are considered good candidates for endoluminal repair of abdominal aortic aneurysms. Patients should be heparinized during the implant procedure such that an activated clotting time of 300 seconds is achieved. During implantation of the TALENT endoluminal stent-graft, the pre-implant CT scan and available angiograms are used together with (on-the-table) digital subtraction angiography (DSA), roadmapping, and angiography for proper implant positioning. The TALENT endoluminal stent-graft endoprosthesis is inserted by delivery catheter and introducer sheath via a surgical cutdown (e.g., external iliac artery, femoral artery) approach. The introducer sheath and delivery catheter containing the stent-graft is inserted over a guidewire and advanced into the aorta and above the aneurysm. With the delivery catheter in the correct position, the push rod is held stationary while the outer sheath is slowly withdrawn. The introducer sheath is then withdrawn further until the stent-graft is completely deployed. The balloon may be inflated along the full length of the implanted device to model the springs against the vessel wall and to unravel possible wrinkles in the graft fabric. After deployment of the stent-graft, angiography is performed to verify implant position and to check for the presence of endoleaks.

Subjects will undergo an evaluation of the TALENT endoluminal stent-graft to determine the safety and efficacy of the device as indicated by the adverse event rate, and to determine the risk factors that are most predictive of a successful outcome when used to exclude abdominal aortic aneurysms that require suprarenal fixation in high risk and low risk patients. Follow-up will be completed at 1, 6, 12, 24, 36, 48, and 60 months. Subject evaluation at 1 month will include a complete Physical Examination, Bilateral ABIs, and a Duplex Ultrasound (if not previously completed at time of discharge). Subject evaluation at 6 months will also include a Complete Physical Examination, Bilateral ABIs, Duplex Ultrasound, and Abdominal X-ray (AP, Lateral, 2 Obliques). Subject evaluation at 12, 24, 36, 48, and 60 months will include a Complete Physical Examination, Bilateral ABIs, Abdominal X-ray (AP, Lateral, 2 Obliques), and Spiral CT scan with and without IV Contrast 2.5mm.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject has a proximal AAA neck (distance between the top of the aneurysm and the renal arteries) ≥ 5 mm.
* Subject has a proximal aortic neck diameter ≥ 14 mm and ≤ 32 mm.
* Subject has an angle between the suprarenal aorta and the aneurysm ≤ 60°.
* Subject has renal arteries ≥ 9 cm from the aortic neck bifurcation.
* Subject has proximal and distal iliac neck diameters ≥ 8 mm and ≤ 24 mm.
* Subject has a distal iliac neck length ≥ 15 mm.
* Subject has signed the informed consent.
* Subject will be available for follow-up at periodic intervals after the procedure.

Exclusion Criteria:

* Subject has a document patent inferior mesenteric artery and an occluded or stenotic celiac and superior mesenteric artery.
* Subject has a lesion that cannot be crossed with a guide wire.
* Subject whose arterial access site cannot accommodate the delivery catheter.
* Subject has no distal vascular bed.
* Subject has systemic infection, or is suspected of having systemic infection.
* Subject has an untreatable bleeding diathesis.
* Subject is not available or is not willing to come back for periodic follow-up (surveillance) after the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2002-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Determine the proportion in whom successful implantation is achieved, as indicated by aneurysm exclusion and graft patency. | At implant, time of discharge, and 1, 6, and 12 months.

SECONDARY OUTCOMES:
Determine the proportion of patients who experience adverse events. | During and after implantation.
Determine the proportion of patients who experience comorbidities and overall mortality rates. | During and after implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Becker GJ, Benenati JF, Zemel G, Sallee DS, Suarez CA, Roeren TK, Katzen BT. Percutaneous placement of a balloon-expandable intraluminal graft for life-threatening subclavian arterial hemorrhage. J Vasc Interv Radiol. 1991 May;2(2):225-9. doi: 10.1016/s1051-0443(91)72286-0. PMID 1799760
- [Background] Bickerstaff LK, Hollier LH, Van Peenen HJ, Melton LJ 3rd, Pairolero PC, Cherry KJ. Abdominal aortic aneurysms: the changing natural history. J Vasc Surg. 1984 Jan;1(1):6-12. PMID 6481873
- [Background] Blum U, Langer M, Spillner G, Mialhe C, Beyersdorf F, Buitrago-Tellez C, Voshage G, Duber C, Schlosser V, Cragg AH. Abdominal aortic aneurysms: preliminary technical and clinical results with transfemoral placement of endovascular self-expanding stent-grafts. Radiology. 1996 Jan;198(1):25-31. doi: 10.1148/radiology.198.1.8539389.
- [Background] Pathology of nonspecific abdominal aortic aneurysm disease. In Current Therapy in Vascular Surgery, 2nd edition, CB Ernst and JC Stanley, eds. B.C. Decker, Philadelphia, PA.
- [Background] Collin J, Araujo L, Walton J, Lindsell D. Oxford screening programme for abdominal aortic aneurysm in men aged 65 to 74 years. Lancet. 1988 Sep 10;2(8611):613-5. doi: 10.1016/s0140-6736(88)90649-6. PMID 2900988
- [Background] Cronenwett JL and LN Samspon. 1995. Aneurysms of the abdominal aorta and iliac arteris. In Current Diagnosis and Treatment in Vascular Surgery, 1st edition, RH Dean, JST Yao and DC Brewster, eds. Appleton and Lange, Norwalk, CT. pp 220-238.
- [Background] Dake MD, Miller DC, Semba CP, Mitchell RS, Walker PJ, Liddell RP. Transluminal placement of endovascular stent-grafts for the treatment of descending thoracic aortic aneurysms. N Engl J Med. 1994 Dec 29;331(26):1729-34. doi: 10.1056/NEJM199412293312601. PMID 7984192
- [Background] DUBOST C, ALLARY M, OECONOMOS N. Resection of an aneurysm of the abdominal aorta: reestablishment of the continuity by a preserved human arterial graft, with result after five months. AMA Arch Surg. 1952 Mar;64(3):405-8. No abstract available. PMID 14894065
- [Background] Geroulakos G, Nicolaides A. Infrarenal abdominal aortic aneurysms less than five centimetres in diameter: the surgeon's dilemma. Eur J Vasc Surg. 1992 Nov;6(6):616-22. doi: 10.1016/s0950-821x(05)80838-2. PMID 1451817
- [Background] Gloviczki P. Ruptured abdominal aortic aneurysms. In Vascular Surgery, 4th edition, Rutherford, RB, ed. Saunders, Philadelphia, PA, chapter 76.
- [Background] Hallett JW Jr, Bower TC, Cherry KJ, Gloviczki P, Joyce JW, Pairolero PC. Selection and preparation of high-risk patients for repair of abdominal aortic aneurysms. Mayo Clin Proc. 1994 Aug;69(8):763-8. doi: 10.1016/s0025-6196(12)61096-9. PMID 8035633
- [Background] Ingoldby CJ, Wujanto R, Mitchell JE. Impact of vascular surgery on community mortality from ruptured aortic aneurysms. Br J Surg. 1986 Jul;73(7):551-3. doi: 10.1002/bjs.1800730711. PMID 3730787
- [Background] Johansson G, Swedenborg J. Ruptured abdominal aortic aneurysms: a study of incidence and mortality. Br J Surg. 1986 Feb;73(2):101-3. doi: 10.1002/bjs.1800730205. PMID 3947894
- [Background] Johansen K. Ruptured abdominal aortic aneurysm: how should recent outcome studies impact current practices? Semin Vasc Surg. 1995 Jun;8(2):163-7. No abstract available. PMID 7670667
- [Background] Johnston KW. Nonruptured abdominal aortic aneurysm: six-year follow-up results from the multicenter prospective Canadian aneurysm study. Canadian Society for Vascular Surgery Aneurysm Study Group. J Vasc Surg. 1994 Aug;20(2):163-70. doi: 10.1016/0741-5214(94)90002-7. PMID 8040938
- [Background] Lee JT, Lee J, Aziz I, Donayre CE, Walot I, Kopchok GE, Heilbron M Jr, Lippmann M, White RA. Stent-graft migration following endovascular repair of aneurysms with large proximal necks: anatomical risk factors and long-term sequelae. J Endovasc Ther. 2002 Oct;9(5):652-64. doi: 10.1177/152660280200900517. PMID 12431151
- [Background] Melton LJ 3rd, Bickerstaff LK, Hollier LH, Van Peenen HJ, Lie JT, Pairolero PC, Cherry KJ, O'Fallon WM. Changing incidence of abdominal aortic aneurysms: a population-based study. Am J Epidemiol. 1984 Sep;120(3):379-86. doi: 10.1093/oxfordjournals.aje.a113902. PMID 6475915
- [Background] Nehler MR, Taylor LM Jr, Moneta GL, Porter JM. Indications for operation for infrarenal abdominal aortic aneurysms: current guidelines. Semin Vasc Surg. 1995 Jun;8(2):108-14. No abstract available. PMID 7670661
- [Background] Nevitt MP, Ballard DJ, Hallett JW Jr. Prognosis of abdominal aortic aneurysms. A population-based study. N Engl J Med. 1989 Oct 12;321(15):1009-14. doi: 10.1056/NEJM198910123211504. PMID 2674715
- [Background] O'Donnell TF, Darling RC, Linton RR. Is 80 years too old for aneurysmectomy? Arch Surg. 1976 Nov;111(11):1250-7. doi: 10.1001/archsurg.1976.01360290084012. PMID 985073
- [Background] O'Hara PJ, Hertzer NR, Krajewski LP, Tan M, Xiong X, Beven EG. Ten-year experience with abdominal aortic aneurysm repair in octogenarians: early results and late outcome. J Vasc Surg. 1995 May;21(5):830-7; discussion 837-8. doi: 10.1016/s0741-5214(05)80015-1. PMID 7769742
- [Background] Pairolero PC. Repair of abdominal aortic aneurysms in high-risk patients. Surg Clin North Am. 1989 Aug;69(4):755-63. doi: 10.1016/s0039-6109(16)44882-6. PMID 2749441
- [Background] Parodi JC, Palmaz JC, Barone HD. Transfemoral intraluminal graft implantation for abdominal aortic aneurysms. Ann Vasc Surg. 1991 Nov;5(6):491-9. doi: 10.1007/BF02015271. PMID 1837729
- [Background] Perler BA. 1995. Natural history of abdominal aortic aneurysm. A clinical presentation. Seventh Annual International Symposium on Vascular Diagnosis and Intervention. pp. 173-175.
- [Background] Rose WM 3rd, Ernst CB. Abdominal aortic aneurysm. Compr Ther. 1995 Jul;21(7):339-43. No abstract available. PMID 7554809
- [Background] Scott RA, Ashton HA, Kay DN. Abdominal aortic aneurysm in 4237 screened patients: prevalence, development and management over 6 years. Br J Surg. 1991 Sep;78(9):1122-5. doi: 10.1002/bjs.1800780929. PMID 1933203
- [Background] Veith FJ, Abbott WM, Yao JS, Goldstone J, White RA, Abel D, Dake MD, Ernest CB, Fogarty TJ, Johnston KW, et al. Guidelines for development and use of transluminally placed endovascular prosthetic grafts in the arterial system. Endovascular Graft Committee. J Vasc Surg. 1995 Apr;21(4):670-85. doi: 10.1016/s0741-5214(95)70198-2. No abstract available. PMID 7707571
- [Background] Zarins CK, Harris EJ Jr. Operative repair for aortic aneurysms: the gold standard. J Endovasc Surg. 1997 Aug;4(3):232-41. doi: 10.1583/1074-6218(1997)0042.0.CO;2. PMID 9291048